CLINICAL TRIAL: NCT04400097
Title: The Influence of Suture Method in Conjunctival Autograft Transplantation on Postoperative Ocular Discomfort for Primary Pterygium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHAIER2020IRB03
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: the Efficacy and Effect on Patient Comfort of a Hidden-knot Continuous Suture for Pterygium Excision With Conjunctival Autograft
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hidden-knot group (Experimental)
  Interventions: Procedure: suture
- two-knot group (Active Comparator)
  Interventions: Procedure: suture
- multi-knot group (Active Comparator)
  Interventions: Procedure: suture

INTERVENTIONS:
Procedure: suture — suture methods of autograft conjunctival transplantation

SUMMARY:
To evaluate the efficacy and effect on patient comfort of a hidden-knot continuous suture for pterygium excision with conjunctival autograft，compared with two-knot continuous sutures and multi-knot interrupted sutures.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary pterygium

Exclusion Criteria:

* eye surgery history
* acute ocular surface imflamation
* patients with coagulation or diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-21 (Estimated); Primary Completion 2020-11-21 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
Patient comfort | 6 months
  discomfort grading on a visual analog scale

IPD SHARING:
Plan to Share IPD: No